CLINICAL TRIAL: NCT05968287
Title: Evaluation of the Relationship of Neutrophil Functions With Sepsis and Septic Shock Using the Leukocyte ImmunoTest™ in Patients With Various Infectious Conditions
Brief Title: Can Measurement of Neutrophil-derived ROS Production be a Novel Biomarker of Sepsis?
Acronym: LIT-sepsis
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Collaborators: Seroxo Ltd (Industry)
Responsible Party: Principal Investigator, Nazlıhan Boyacı Dündar, assistan professor, Division of Intensive Care Medicine (principle invastigator), Gazi University
Other Study IDs: GaziUtipNBDundar002
Record Dates: First submitted 2023-07-04; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Infections; Sepsis; Septic Shock
Keywords: cellular dysfunction of neutrophils; reactive oxygen species (ROS); sepsis; septic shock; infections; biomarker
MeSH Terms: conditions — Infections; Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patient group: patients admitted to hospital with various infection conditions with or without sepsis
  Interventions: Diagnostic Test: The Leukocyte ImmunoTest™ (LIT™)
- control group: patients admitted to hospital with various non-infectious diseases and outpatients who admitted to the outpatient clinics
  Interventions: Diagnostic Test: The Leukocyte ImmunoTest™ (LIT™)

INTERVENTIONS:
Diagnostic Test: The Leukocyte ImmunoTest™ (LIT™) — The baseline LIT scores was performed for two parallel groups. The sequential LIT score was also performed for patients with various infection conditions with/without sepsis.

SUMMARY:
Neutrophils are indispensable for host defense and have an important roles in modulating the immune system in both the innate and adaptive immune response. Neutrophils operate using a number of different mechanisms including chemotaxis, phagocytosis, release of reactive oxygen species (ROS) and granular proteins, and the production and liberation of cytokines for this purpose. A controlled neutrophil response is required to combat infection; an dysregulated state of this response can cause sepsis, tissue damage, and organ failure. Sepsis and septic shock are the leading causes of death especially in intensive care units (ICU), and their mortality can be reduced with prompt diagnosis and appropriate treatment modality. From this point of view, many biomarkers have been evaluated for the diagnosis, prognosis, and treatment response of infection and sepsis. An objective marker of cellular dysfunction of neutrophils would be a helpful tool for the clinician in detecting and monitoring changes related to infection status and to determine development of sepsis and positive effects of interventions.

DETAILED DESCRIPTION:
Introduction:

Sepsis is defined as the dysregulated host response to infection leading to organ dysfunction. Both sepsis and septic shock are important health problems affecting millions of people, resulting in a serious mortality rate around the world every year. Delay in both diagnosis and initiation of appropriate treatment are the most important causes of sepsis-related mortality. On the other hand, overdiagnosis of sepsis and initiation of broad-spectrum antibiotic therapy inappropriately have some consequences such as increased hospital costs, antibiotic-related side effects, increased antibiotic resistance, and the development of resistant nosocomial infections. To make this precise distinction, a large number of biomarkers have been studied until today. The expected benefit of sepsis-related biomarkers is the detection of infection and sepsis, the potential to predict the course of sepsis, or treatment guidance. Although there are more than 150 biomarkers studied on this subject, there is not a single biomarker that meets these expectations in all aspects in clinical practice.

Neutrophils play a vital role in the development of the host response in sepsis. Neutrophils operate using a number of different mechanisms including chemotaxis, phagocytosis, release of reactive oxygen species (ROS) and granular proteins, and the production and liberation of cytokines for this purpose. A controlled neutrophil response is required to combat infections. Recently a functional assay that assesses the capacity of leukocytes (primarily neutrophils) to produce ROS in response to in vitro chemical stimulation has been demonstrated. The Leukocyte ImmunoTest™ (LIT™) specifically and rapidly (10 minutes) quantifies neutrophil ROS release using a small volume of blood obtainable from capillary, arterial or venous sources. As such the LIT score provides a physiologically relevant means for monitoring the cellular capacity of neutrophils to produce superoxide radicals in real time. An objective marker of cellular dysfunction of neutrophils would be a helpful tool for the clinician in detecting and monitoring changes related to infection status and to determine development of sepsis and positive effects of interventions.

Method:

The study was conducted as a prospective observational study with ethical committee approval in a medical intensive care unit and inward belong to internal disease department of a university hospital. The patient population is consisted of patients who were admitted to the ICU or inward due various infectious etiologies. The control group is consisted of outpatients or inpatients admitted to ICU or inward for noninfectious etiologies. ROS production in response to PMA was performed on clinical samples and analysed within 30 minutes of collection. The LIT test was performed every day or every other day for patient group until death or discharge from units where the study is conducted. The LIT test was performed only once for outpatient group on day of outpatient control.

Measurements of ROS production by luminometer:

ROS production was measured on clinical samples taken for routine testing. Briefly, 10μl samples of freshly obtained blood (obtained by venepuncture) was added to 100 microlitres phosphate buffered saline (PBS) containing phorbol 12-myristate 13-acetate (PMA; Sigma) and luminol. The solution was incubated for 10 minutes at 37.5 °C. Chemiluminescence was quantified after 10 minutes using handheld luminometer (3M, Clean-Trace, NG3) in relative light units (RLU). LIT scores as a correlate of neutrophil function for each patient were plotted. Abnormally high (hyperproduction) ROS generation was associated with infection, sepsis or septic shock. This raises the possibility of LIT™ and LIT™/neutrophil-count ratio, (LIT/N), being used as a predictive clinical tool.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis or suspicion of various infectious disease with or without sepsis and admitted to the ICU or inpatient service due to this clinical diagnosis for patient group
2. Patients followed in the inpatient service due to various non-infectious diseases and outpatients who were examined in outpatient clinics for control group

Exclusion Criteria:

1. patient or control group under the age of 18 years
2. Patients died within the 24 hours after hospital admission
3. Patients who did not sign informed consent
4. Refusal of legal representative to participate in the study in unconscious patients
5. Patients with an absolute neutrophil count <500/mm3 on admission
6. Control group describing any infective symptoms
7. Control group with a chronic infectious disease under treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population is consisted of patients who were admitted to the ICU or inward due various infectious etiologies. The control population is consisted of outpatients or inpatients admitted to ICU or inward for noninfectious etiologies.
Sampling Method: Non-Probability Sample
Enrollment: 276 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
the reactive oxygen species (ROS) production of neutrophils via the Leukocyte ImmunoTest™ (LIT) | Patients' LIT scores in relative light units (RLU) within 24 hours following the day of hospitalization during the study period
  the difference of the Leukocyte ImmunoTest™ (LIT) as relative light unit (RLU) between patients with various infection conditions and control groups without infection.
  Abnormally high (hyperproduction) ROS generation demonstrated via The Leukocyte ImmunoTest™ (LIT) is associated with infection. LIT scores as relative light unit (RLU) can vary between 1-15000.
the reactive oxygen species (ROS) production of neutrophils via the Leukocyte ImmunoTest™ (LIT) | LIT score as as relative light unit (RLU) of the day of detecting of infection and sepsis up to 8 months
  the difference of the Leukocyte ImmunoTest™ (LIT) as relative light unit (RLU) between patients between sepsis and without sepsis
  Abnormally high (hyperproduction) ROS generation demonstrated via The Leukocyte ImmunoTest™ (LIT) is associated with sepsis and septic shock. LIT scores as relative light unit (RLU) can vary between 1-15000.

SECONDARY OUTCOMES:
the reactive oxygen species (ROS) production of neutrophils via the Leukocyte ImmunoTest™ (LIT) | the Leukocyte ImmunoTest™ (LIT) as relative light unit (RLU) of the patients with sepsis on every day or every other day up to death or discharge from the hospital through the study completion, an average of 8 months
  the difference of the Leukocyte ImmunoTest™ (LIT) as relative light unit (RLU) between survivors and nonsurvivors within the septic patients.
  Abnormally high (hyperproduction) ROS generation demonstrated via The Leukocyte ImmunoTest™ (LIT) is associated with infection, sepsis and septic shock. LIT scores as relative light unit (RLU) can vary between 1-15000. The relationship of high scores of the LIT as relative light unit (RLU) with mortality will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Nazlıhan Boyacı Dündar, assist.prof., Principal Investigator — principle investigator
Locations (1):
- Gazi University, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mortaz E, Alipoor SD, Adcock IM, Mumby S, Koenderman L. Update on Neutrophil Function in Severe Inflammation. Front Immunol. 2018 Oct 2;9:2171. doi: 10.3389/fimmu.2018.02171. eCollection 2018. PMID 30356867
- [Background] Selders GS, Fetz AE, Radic MZ, Bowlin GL. An overview of the role of neutrophils in innate immunity, inflammation and host-biomaterial integration. Regen Biomater. 2017 Feb;4(1):55-68. doi: 10.1093/rb/rbw041. PMID 28149530
- [Background] Hellebrekers P, Vrisekoop N, Koenderman L. Neutrophil phenotypes in health and disease. Eur J Clin Invest. 2018 Nov;48 Suppl 2(Suppl Suppl 2):e12943. doi: 10.1111/eci.12943. Epub 2018 May 25. PMID 29682724
- [Background] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Moller MH, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving sepsis campaign: international guidelines for management of sepsis and septic shock 2021. Intensive Care Med. 2021 Nov;47(11):1181-1247. doi: 10.1007/s00134-021-06506-y. Epub 2021 Oct 2. No abstract available. PMID 34599691
- [Background] Ferrer R, Martin-Loeches I, Phillips G, Osborn TM, Townsend S, Dellinger RP, Artigas A, Schorr C, Levy MM. Empiric antibiotic treatment reduces mortality in severe sepsis and septic shock from the first hour: results from a guideline-based performance improvement program. Crit Care Med. 2014 Aug;42(8):1749-55. doi: 10.1097/CCM.0000000000000330. PMID 24717459
- [Background] Pierrakos C, Velissaris D, Bisdorff M, Marshall JC, Vincent JL. Biomarkers of sepsis: time for a reappraisal. Crit Care. 2020 Jun 5;24(1):287. doi: 10.1186/s13054-020-02993-5. PMID 32503670
- [Background] Fleischmann-Struzek C, Mellhammar L, Rose N, Cassini A, Rudd KE, Schlattmann P, Allegranzi B, Reinhart K. Incidence and mortality of hospital- and ICU-treated sepsis: results from an updated and expanded systematic review and meta-analysis. Intensive Care Med. 2020 Aug;46(8):1552-1562. doi: 10.1007/s00134-020-06151-x. Epub 2020 Jun 22. PMID 32572531
- [Background] Rhee C, Chiotos K, Cosgrove SE, Heil EL, Kadri SS, Kalil AC, Gilbert DN, Masur H, Septimus EJ, Sweeney DA, Strich JR, Winslow DL, Klompas M. Infectious Diseases Society of America Position Paper: Recommended Revisions to the National Severe Sepsis and Septic Shock Early Management Bundle (SEP-1) Sepsis Quality Measure. Clin Infect Dis. 2021 Feb 16;72(4):541-552. doi: 10.1093/cid/ciaa059. PMID 32374861
- [Background] Biomarkers Definitions Working Group.. Biomarkers and surrogate endpoints: preferred definitions and conceptual framework. Clin Pharmacol Ther. 2001 Mar;69(3):89-95. doi: 10.1067/mcp.2001.113989. No abstract available. PMID 11240971
- [Background] Veenith T, Martin H, Le Breuilly M, Whitehouse T, Gao-Smith F, Duggal N, Lord JM, Mian R, Sarphie D, Moss P. High generation of reactive oxygen species from neutrophils in patients with severe COVID-19. Sci Rep. 2022 Jun 21;12(1):10484. doi: 10.1038/s41598-022-13825-7. PMID 35729319
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338